CLINICAL TRIAL: NCT06685536
Title: A Long-term Follow-up Study Evaluating the Safety and Efficacy of Subjects With β-thalassemia Treated With Base-edited Autologous Hematopoietic Stem Cell (CS-101) Transplantation
Brief Title: A Long-term Follow-up Study in Participants Who Received CS-101
Status: Enrolling by invitation | Type: Observational
Sponsor: CorrectSequence Therapeutics Co., Ltd (Industry)
Collaborators: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: CS-101-13
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia | interventions — Safety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Safety and efficacy assessments — Safety evaluations,disease-specific assessments,and assessments to monitor for long-term complications of autologous transplant

SUMMARY:
This is a study to evaluate the long-term safety and efficacy of CS-101 in participants who received CS-101 in study CS -101-06 (NCT06024876),No investigational drug product will be administered in the study.

DETAILED DESCRIPTION:
This is a study to evaluate the long-term safety and efficacy of CS-101 in participants who received CS-101 in study CS -101-06 (NCT06024876). Subjects in the CS-101-06 study will be entered into long-term follow-up of this study up to 15 years post-infusion at the completion of the last (12-month) followup visit after treatment with CS-101 Injection.

ELIGIBILITY:
Inclusion Criteria:

* Participants (or his or her legally appointed and authorized representative or guardian) must sign and date informed consent form (ICF) and, where applicable, an assent form
* Participants must have received CS-101 infusion in last study

Exclusion Criteria:

* There are no exclusion criteria

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subject with β-thalassemia treated with CS-101 infusion in last study
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2025-01-18 (Actual); Primary Completion 2039-07 (Estimated); Study Completion 2039-07 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of SAEs and CS-101 related AES as assessed by CTCAE v5.0 | Through 15 years post CS-101 infusion
  CommonTerminology Criteria for Adverse Events#CTCAE#has 5 levels of AE determination, increasing in severity as the level increases
New malignancies and hematologic disorders | Through 15 years post CS-101 infusion
  Based on ICD-11
Occurrence of all-cause death | Through 15 years post CS-101 infusion
Occurrence of achieving transfusion independence for at least 12 consecutive months | Through 15 years post CS-101 infusion

SECONDARY OUTCOMES:
Change in fetal hemoglobin(HbF) concentration over time | Through 15 years post CS-101 infusion
Change in total hemoglobin(Hb) concentration over time | Through 15 years post CS-101 infusion
Chimerism level in Peripheral blood Proportion of alleles with intended genetic modification in | Through 15 years post CS-101 infusion
Chimerism level in bone marrow Proportion of alleles with intended genetic modification in | Through 15 years post CS-101 infusion
Change in F-Cell concentration over time | Through 15 years post CS-101 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Yongrong Lai, M.D., Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No